CLINICAL TRIAL: NCT04742387
Title: Assessment of Bone Mineral Density in People Living With HIV and KSHV Associated Malignancies: A Retrospective Longitudinal Analysis
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000265; 000265-C
Record Dates: First submitted 2021-02-05; First posted 2021-02-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: Kaposi Sarcoma; KSHV Associated Multicentric Castleman Disease; Primary Effusion Lymphoma; IL-6 Related KSHV Associated Cytokine Syndrome
Keywords: AIDS; Antiretroviral Therapy; OSTEOPENIA; bone turnover markers; Natural History
MeSH Terms: conditions — Sarcoma, Kaposi; Multi-centric Castleman's Disease; Lymphoma, Primary Effusion; Acquired Immunodeficiency Syndrome; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Medical records of subjects enrolled on various studies conducted by HAMB/CCR from 1/1/2005 to 12/1/2020

SUMMARY:
Background:

Some people with human immunodeficiency virus (HIV) are on antiretroviral therapy (ART). Their cells have shown to age faster than expected. This puts them at higher risk for a range of age-related diseases about 10 years sooner than people who do not have HIV. Low bone mineral density (BMD) is common in people with HIV. This means their risk of fractures is increased. People with HIV also have a higher risk for cancers caused by Kaposi's sarcoma herpesvirus (KSHV) than people who do not have HIV. Much of the data on bone loss related to cancer and cancer treatments has been gathered from people who do not have HIV. Researchers want to learn more about the rate of bone loss in people with HIV/AIDS and KSHV associated cancers.

Objective:

To learn the factors that are linked to BMD loss in people with HIV and KSHV associated cancers from imaging performed as part of NIH studies.

Eligibility:

Adults with HIV and Kaposi s sarcoma who got ART and cancer chemotherapy at NIH from 1/1/2005 to 12/1/2020.

Design:

Participants' records will be chosen from studies that were conducted from 1/1/2005 to 12/1/2020. This study will include participants who had at least 2 CT scans. Some participants may have opted out of the future use of their data. If so, their records will not be used.

This study will use data collected at NIH. Data taken from CT scans will be used to measure BMD.

Study results may be published.

This study will last about 2 years.

DETAILED DESCRIPTION:
Title:

Assessment of Bone Mineral Density in People Living with HIV and KSHV Associated Malignancies: A Retrospective Longitudinal Analysis

Study Description:

This is a retrospective review that includes all participants with human immunodeficiency virus (HIV) (PWH) affected by Kaposi sarcoma (KS), KSHV-associated multicentric Castleman disease, and KSHV associated inflammatory cytokine syndrome enrolled on the tissue procurement study (01-C-0038) and other treatment protocols within the HIV/AIDS Malignancy Branch at the National Cancer Institute (NCI) from 1/1/2005 to 12/1/2020.

Objectives:

To determine the factors that are associated with bone mineral density (BMD) loss in PWH and KSHV associated malignancies.

Study Population:

All patients seen at the NIH from 1/1/2005 to 12/1/2020.

Description of Sites/Facilities conducting research:

This is a single site study initiated by the HIV/AIDS Malignancy Branch at the National Cancer Institute

Study Duration:

Data abstraction to completion of data analyses will take about 2 years.

ELIGIBILITY:
* STUDY POPULATION:

Subjects will not be recruited for this study; however, participants' records will be selected from treatment protocols from 1/1/2005 to 12/1/2020 unless the subject opted out of the future use of his/her data. These subjects enrolled to natural history and/or treatment protocols within the HIV/AIDS Malignancy Branch on the basis of a diagnosis of HIV and KSHV-associated conditions, such as KS alone, in combination with KSHV-MCD or KICS.

As this is a retrospective longitudinal study, the investigators will review the data from subjects who have at least two completed CT scans to measure bone mineral density.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
BMD loss | ongoing
  To determine variables that are associated with BMD loss in participants with HIV and KSHV associated malignancies from retrospective imaging performed as part of clinical research protocols

SECONDARY OUTCOMES:
longitudinal change in BMD | ongoing
  To estimate the longitudinal change in BMD from study baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ramya M Ramaswami, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States